CLINICAL TRIAL: NCT04984343
Title: Randomized Phase II Trial of Five or Two MRI-Guided Adaptive Radiotherapy Treatments for Prostate Cancer
Brief Title: Randomized Trial of Five or Two MRI-Guided Adaptive Radiotherapy Treatments for Prostate Cancer
Acronym: FORT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Viewray Inc. (Industry); Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-02023315
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Low or intermediate risk prostate cancer; Definitive radiotherapy; MRI Linear accelerator
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 5 radiation treatments - ARM 1 (Experimental): Patients randomized to ARM 1 will receive 37.5 in 5 radiotherapy treatments.
  Interventions: Radiation: Radiation Therapy
- 2 radiation treatments - ARM 2 (Active Comparator): Patients randomized to ARM 2 will receive 25 Gy in 2 radiotherapy treatments.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Eligible subjects will be randomly assigned to 5 or 2 fraction treatment groups in a 1:1 ratio using a computer-generated randomization scheme.
  After consent and eligibility verification, patients will undergo CT/MRI simulation and radiotherapy planning. Patients will receive treatment to the prostate +/- seminal vesicles per treating physician's discretion in either 37.5 Gy in 5 fractions or 25 Gy in 2 fractions. SIB use is at treating physician's discretion and should be concordant with imaging and biopsy findings with no PTV expansion.
  Subjects on 5 fraction arm should be treated on non-consecutive days. Subjects on the 2 fraction arm must have >72 hours between beginning of each fraction.

SUMMARY:
The study is a randomized study that compares 5 radiation therapy treatments to 2 radiation therapy treatments in men with low or intermediate-risk prostate cancer.

DETAILED DESCRIPTION:
This study is a randomized non-inferiority trial comparing 5 to 2 radiotherapy treatments using an MRI linear accelerator for men with low or intermediate-risk prostate cancer electing for definitive radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Men aged >=18 with histologically confirmed low or intermediate risk prostate cancer per NCCN guidelines.
* ECOG 0 - 1
* IPSS < 18
* Ability to receive MRI-guided radiotherapy.
* Ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire.
* Patients with a prior or concurrent disease whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Note: Any patient with a cancer (other than keratinocyte carcinoma or carcinoma in situ or low-grade non-muscle invasive bladder cancer) who has been disease-free for less than 3 years must contact the Principal Investigator.

Exclusion Criteria:

* Prior history of receiving pelvic radiotherapy.
* Patient with history of inflammatory bowel disease.
* MRI Prostate Volume > 80 cc
* MRI Stage > T3a
* Unilateral or bilateral hip replacements.
* History of bladder neck or urethral stricture.
* TURP < 8 weeks prior to radiotherapy
* Metastatic (pelvic nodal or distant) disease on CT, Bone, Fluciclovine, and/or PSMA PET scan

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of patient-reported GI symptoms using the Expanded Prostate Cancer Index Composite (EPIC) | Baseline, 24 months
  The primary objective is to demonstrate that 2 treatments of radiotherapy does not significantly increase patient-reported Gastrointestinal (GI) and Genitourinary (GU) symptoms compared to 5 treatments of radiotherapy 2 years after treatment completion.

SECONDARY OUTCOMES:
Change in the number of patient reported GI symptoms at specific intervals as measured by Expanded Prostate Cancer Index Composite (EPIC) | Baseline, 1 week , 3months, 6 months, 12 months and 60 months
  Compare patient-reported GI symptoms using the EPIC at end of RT and 3, 6, 12, and 60 months from end of treatment.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
  Adverse events can be unexpected or expected, related to treatment.
Change in the number of patient reported GU symptoms at specific intervals as measured by Expanded Prostate Cancer Index Composite (EPIC) | Baseline, 1 week, 3months, 6 months, 12 months and 60 months
  Compare patient-reported GU symptoms using the EPIC at end of RT and 3, 6, 12, and 60 months from end of treatment.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
  Adverse events can be unexpected or expected, related to treatment.
Change in the number of patient reported sexual symptoms at specific intervals as measured by Expanded Prostate Cancer Index Composite (EPIC) | Baseline, 1 week, 3months, 6 months, 12 months and 60 months
  Compare patient-reported sexual symptoms using the EPIC at end of RT and 3, 6, 12, 24, and 60 months from end of treatment.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
  Adverse events can be unexpected or expected, related to treatment.
Time to Progression (TTP) | 3 months
  Compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (PCSM).
Time to Progression (TTP) | 6 months
  Compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (PCSM).
Time to Progression (TTP) | 12 months
  Compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (PCSM).
Time to Progression (TTP) | 60 months
  Compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (PCSM).
Compare Overall Survival Rates | 3 months
  Compare Overall Survival (OS) in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
Compare Overall Survival Rates | 6 months
  Compare Overall Survival (OS) in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
Compare Overall Survival Rates | 12 months
  Compare Overall Survival (OS) in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
Compare Overall Survival Rates | 60 months
  Compare Overall Survival (OS) in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
prostate cancer specific survival | 3 months
  compare prostate cancer specific survival in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
prostate cancer specific survival | 6 months
  compare prostate cancer specific survival in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
prostate cancer specific survival | 12 months
  compare prostate cancer specific survival in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.
prostate cancer specific survival | 60 months
  compare prostate cancer specific survival in patients among the two arms, 37.5 Gy in 5 fractions and 25 Gy in 2 fractions.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Weg, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- Weill Cornell Medicine, New York, New York, United States
- Genesis Care, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolfe S, Diven MA, Marciscano AE, Zhou XK, Kishan AU, Steinberg ML, Miccio JA, Camilleri P, Nagar H. A randomized phase II trial of MR-guided prostate stereotactic body radiotherapy administered in 5 or 2 fractions for localized prostate cancer (FORT). BMC Cancer. 2023 Sep 30;23(1):923. doi: 10.1186/s12885-023-11430-z. PMID 37777738